CLINICAL TRIAL: NCT01570231
Title: Feasibility, Safety and Efficacy of RIPC for Symptomatic Intracranial Arterial Stenosis in Octogenarians
Brief Title: Feasibility, Safety and Efficacy of Remote Ischemic Preconditioning for Symptomatic Intracranial Arterial Stenosis in Octogenarians
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ji Xunming (Other)
Collaborators: Capital Medical University (Other)
Responsible Party: Sponsor-Investigator, Ji Xunming, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2009
Record Dates: First submitted 2012-03-25; First posted 2012-04-04 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Bilateral Limb Ischemic Preconditioning; Intracranial Arterial Stenosis
Keywords: remote ischemic preconditioning; octogenarian; intracranial arterial stenosis; stroke recurrence

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- bilateral limb ischemic preconditioning (BLIPC) (Experimental): 5 minutes bilateral limb ischemic preconditioning treatment with an inflating tourniquets to 200 mmHg
  Interventions: Device: bilateral limb ischemic preconditioning (Doctormate, IPC-906X)
- Control group (No Intervention): underwent equivalent medical treatments only

INTERVENTIONS:
Device: bilateral limb ischemic preconditioning (Doctormate, IPC-906X) — Device: bilateral limb ischemic preconditioning (Doctormate, IPC-906X, produced by Beijing Renqiao Institute of Neuroscience)five cycles of 5 minutes bilateral upper limb ischemia-reperfusion performed by inflating tourniquets to 200 mmHg, twice daily for 180 consecutive days, along with conventional medical treatment.
  Arms: bilateral limb ischemic preconditioning (BLIPC)

SUMMARY:
Making a limb transiently ischemic induces ischemic tolerance in distant organs such as the heart. This study aims to evaluate the feasibility, safety and initial efficacy of using briefly repetitive bilateral limb ischemic preconditioning (BLIPC) to protect the brain in octogenarians with symptomatic intracranial arterial stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. age between 80 to 95 years old
2. Trial of Org 10172 in Acute Stroke Treatment-1 (TOAST-1) subtype
3. National Institutes of Health Stroke Scale (NIHSS) score 0-15, and Modified Rankin Scale (mRS) score 0-4
4. ABCD2 score between 6 to 7
5. stable vital signs, normal hepatic and renal functions
6. no hemorrhagic tendencies

Exclusion Criteria:

1. within 72 hrs of intra-artery or intravenous thrombolysis
2. intracranial hemorrhage or large area of cerebral infarction (more than 1/3 middle cerebral artery perfusion territory)
3. any soft tissue, orthopedic, or vascular injury, wounds or fractures in extremities which may pose a contraindication for application of the preconditioning cuffs
4. acute myocardial infarction
5. systolic blood pressure more than 200 mmHg after drug control
6. peripheral blood vessel disease
7. hematologic disease
8. severe hepatic and renal dysfunction
9. severe or unstable concomitant disease
10. cannot tolerate BLIPC or without informed consent

Ages: 80 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
objective signs of tissue or neurovascular injury | 180 days after treatment
  objective signs of tissue or neurovascular injury felt to be due to cuff inflation, which was based on the judgment of the observers (blinded to study protocol) precluded continuation. Inspection included palpation of distal radial pulses, visual inspection (for local edema, redness, skin breakdown), and palpation for tenderness
levels of plasma biomarkers | 180-day
  levels of plasma myoglobin at baseline and at the 1st, 15th and 30th day during BLIPC treatment were monitored

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Meng R, Ding Y, Asmaro K, Brogan D, Meng L, Sui M, Shi J, Duan Y, Sun Z, Yu Y, Jia J, Ji X. Ischemic Conditioning Is Safe and Effective for Octo- and Nonagenarians in Stroke Prevention and Treatment. Neurotherapeutics. 2015 Jul;12(3):667-77. doi: 10.1007/s13311-015-0358-6. PMID 25956401